CLINICAL TRIAL: NCT05274178
Title: Effect of Hearing Aid Labeling on Speech Understanding Measures
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Sonova AG (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Crossover | Masking: Single | Purpose: Treatment
Other Study IDs: SRF-505
Record Dates: First submitted 2022-03-01; First posted 2022-03-10 (Actual); Results first posted 2023-07-10 (Actual); Last update posted 2023-07-10 (Actual); Status verified 2023-06

CONDITIONS: Hearing Loss
MeSH Terms: conditions — Hearing Loss

STUDY DESIGN:
Intervention Model Description: A single group of participants will be involved in this study. All participants will be evaluated with both hearing devices.
Who Masked: Investigator
Masking Description: Participants will be told they are wearing either a prescriptive hearing aid or an OTC (Over-The-Counter) hearing device based on the labeling of the hearing aids. Both sets of devices will actually be the same. The investigator that is scoring the objective speech in noise test will not know which device the participant is wearing at the time of the test (i.e., the set that is labeled as prescriptive or the set that is labeled as OTC).
Oversight: FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: Yes

ARMS (2):
- Naive listeners (Experimental): Participants who have never worn a hearing aid before. This group will be tested with both sets of devices, those labeled as "OTC" and those labeled as "Prescriptive"
  Interventions: Device: Audeo P hearing aid labeled as "Prescriptive"; Device: Audeo P hearing aid labeled as "OTC"
- Experienced users (Experimental): Participants who have at least six months experience wearing hearing aids. This group will be tested with both sets of devices, those labeled as "OTC", and those labeled as "Prescriptive"
  Interventions: Device: Audeo P hearing aid labeled as "Prescriptive"; Device: Audeo P hearing aid labeled as "OTC"

INTERVENTIONS:
Device: Audeo P hearing aid labeled as "Prescriptive" — The Audeo P is a commercially available hearing aid that is fit by a hearing care professional. The devices will be labeled as "prescriptive" in view of the participant.
Device: Audeo P hearing aid labeled as "OTC" — The Audeo P is a commercially available hearing aid that is fit by a hearing care professional. The devices will be labeled as "OTC" in view of the participant.

SUMMARY:
New and experienced hearing aid users will be fit with two hearing devices. One will be labeled as an OTC (Over-The-Counter) device, the other will be labeled as a Prescriptive (i.e. professionally fit) device. Both devices will be generically programmed for a mild to moderate hearing loss. An objective speech in noise test will be completed with both devices.

ELIGIBILITY:
Inclusion Criteria:

* Adults age 18 or older with bilateral mild to moderate hearing loss
* Experienced users must have at least 6 months Hearing Aid experience
* New users must have no prior hearing aid experience, defined as never owning their own devices

Exclusion Criteria:

* Self-reported ear related pathology (otorrhea w/in 90 days, dizziness, sudden hearing loss or worsening of hearing w/in 90 days, otalgia)
* Visible deformity of the ear
* Chronic, severe tinnitus
* Unilateral hearing loss
* Cognitive impairment

Ages: 18 Years to 95 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 20 (Actual)
Dates: Start 2022-05-26 (Actual); Primary Completion 2022-06-16 (Actual); Study Completion 2022-06-16 (Actual)

CONTACTS AND LOCATIONS:
Locations (1):
- Sonova US, Aurora, Illinois, United States

RESULTS

PARTICIPANT FLOW:
Groups:
- Naive Listeners: Participants who have not worn hearing aids before. These participants will be tested with both sets of Audeo P hearing aids. One set will be labeled as "OTC" and the other set will be labeled as "Prescriptive".
  Audeo P hearing aid labeled as "Prescriptive": The Audeo P is a commercially available hearing aid that is fit by a hearing care professional. The devices will be labeled as "prescriptive" in view of the participant.
  Audeo P hearing aid labeled as "OTC": The Audeo P is a commercially available hearing aid that is fit by a hearing care professional. The devices will be labeled as "OTC" in view of the participant.
- Experienced Users: Participants who have at least 6 months experience with hearing aids. These participants will be tested with both sets of Audeo P hearing aids. One set will be labeled as "OTC" and the other set will be labeled as "Prescriptive".
  Audeo P hearing aid labeled as "Prescriptive": The Audeo P is a commercially available hearing aid that is fit by a hearing care professional. The devices will be labeled as "prescriptive" in view of the participant.
  Audeo P hearing aid labeled as "OTC": The Audeo P is a commercially available hearing aid that is fit by a hearing care professional. The devices will be labeled as "OTC" in view of the participant.
Period: Overall Study
Arm/Group | Naive Listeners | Experienced Users
Started | 10 | 10
Tested With "OTC" Labeled Devices | 10 | 10
Tested With "Prescriptive" Laeled Devices | 10 | 10
Completed | 10 | 10
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Experienced Users: Participants who haveat least 6 months of experience with hearing aids. These participants will be tested with both sets of Audeo P hearing aids. One set will be labeled as "OTC" and the other set will be labeled as "Prescriptive".
  Audeo P hearing aid labeled as "Prescriptive": The Audeo P is a commercially available hearing aid that is fit by a hearing care professional. The devices will be labeled as "prescriptive" in view of the participant.
  Audeo P hearing aid labeled as "OTC": The Audeo P is a commercially available hearing aid that is fit by a hearing care professional. The devices will be labeled as "OTC" in view of the participant.
- Total: Total of all reporting groups
Arm/Group | Naive Listeners | Experienced Users | Total
Number analyzed (Participants) | 10 | 10 | 20
Age, Continuous [Mean (Full Range); unit: years] | 70 [56 to 81] | 76.8 [69 to 85] | 73.4 [56 to 85]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 7 | 7 | 14
  Male | 3 | 3 | 6
Race and Ethnicity Not Collected [Count of Participants; unit: Participants] — Population: Race and Ethnicity were not collected from any participant.
Region of Enrollment [Number; unit: participants]
  United States | 10 | 10 | 20

OUTCOME MEASURES:

1. Primary Outcome: Quick Speech in Noise Test (QuickSIN)
Description: A speech in noise test in which participant repeats sentences in variable levels of background noise. Test result is reported as the signal to noise level at which participant can repeat 50% of the words correctly. A lower score/dB SNR (decibel Signal to Noise Ratio) level indicates better speech in noise perception. For example, a score of 0 dB would indicate that the participant can repeat 50% of the words presented when the speech signal and the noise are presented at the same level. A score of 6 dB would indicate that the participant needs the speech signal 6 dB louder than the noise in order to correctly repeat 50% of the words presented. Scores can range from negative db SNR (e.g. -5 dB, which would be a good score and indicate little difficulty in noise) to quite high (e.g. +15 dB, which would be a poorer score and indicate much difficulty in noise) In this case, the scores ranged from +2 to +18 dB.
Time Frame: Day 1 of 1 day study
Population: All participants who were tested with the devices labeled as "OTC" and with devices that were labeled as "Prescriptive" in the same test session.
Measure: Mean (Full Range); unit: decibels (dB)
Arm/Group | Naive Listeners | Experienced Users
Number analyzed (Participants) | 10 | 10
decibels (dB)
  dB SNR with "OTC" labelled devices | 6.2 [2 to 12] | 9.6 [3 to 15]
  dB SNR with "Prescriptive" labelled devices | 5.2 [1 to 11] | 10 [2 to 18]
Statistical Analysis 1: Comparison: Naive Listeners; Test type: Other; p > .05, t-test, 2 sided
Statistical Analysis 2: Comparison: Experienced Users; Test type: Other; p > .05, t-test, 2 sided

ADVERSE EVENTS:
Time Frame: 1 day
Arm/Group | Naive Listeners | Experienced Users
All-Cause Mortality (participants affected / at risk) | 0/10 | 0/10
Serious Adverse Events (participants affected / at risk) | 0/10 | 0/10
Other Adverse Events (participants affected / at risk) | 0/10 | 0/10

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2022-05-23): https://cdn.clinicaltrials.gov/large-docs/78/NCT05274178/Prot_SAP_000.pdf